CLINICAL TRIAL: NCT03479697
Title: High-Resolution, Relational, Resonance-Based, Electroencephalic Mirroring (HIRREM) for Stage 1 Primary Hypertension
Brief Title: HIRREM for Stage 1 Primary Hypertension
Acronym: HIRREM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00047477
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2022-07

CONDITIONS: Hypertension; Blood Pressure; Cardiovascular Diseases; Cardiovascular Risk Factor; Autonomic Nervous System Imbalance
Keywords: HIRREM; Neurotechnology; Closed-Loop; Allostasis; Stress; Autonomic Dysregulation; Hyperarousal; Brain Electrical Activity; Acoustic Stimulation; Primary Hypertension; High Blood Pressure
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Primary Dysautonomias; Essential Hypertension

STUDY DESIGN:
Intervention Model Description: This study will compare acoustic stimulation linked to brainwave activity (HIRREM, along with continued current care, HCC), with continued current clinical care alone (CCC). Both groups will continue their other current care throughout, including non-pharmacological, and lifestyle modification therapies. The participants in the CCC group will be offered the opportunity to crossover and receive a course of HCC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- HIRREM (Active Comparator): High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM) is a novel, noninvasive, closed-loop, brainwave mirroring, acoustic stimulation neurotechnology to support relaxation and auto-calibration of neural oscillations, using auditory tones to reflect brain frequencies in near real time.
  Interventions: Device: HIRREM; Other: Continued Current Care
- Continued Current Care (Other): Participants will continue their current care.
  Interventions: Device: HIRREM; Other: Continued Current Care

INTERVENTIONS:
Device: HIRREM — Technology
  Other Names: High-resolution, relational, resonance-based, electroencephalic mirroring; Brainwave Optimization
Other: Continued Current Care — Continue their current clinical care.

SUMMARY:
The purpose of this study is to determine that effects of an intervention called High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM), on Stage 1 Primary Hypertension (systolic BP 130-139, and/or diastolic BP 80-89).

DETAILED DESCRIPTION:
The purpose of this research study is to determine the effects of a technique called High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM®), for hypertension. HIRREM uses scalp sensors to monitor brain electrical activity, and computer software algorithms translate selected brain frequencies into audible tones in real time. Those tones are reflected back to participants via ear buds in as little as four to eight milliseconds, providing the brain an opportunity for self-adjustment of its electrical pattern.

This study will compare acoustic stimulation linked to brainwave activity (HIRREM, along with continued current care, HCC), with continued current clinical care alone (CCC). Both groups will continue their other current care throughout, including non-pharmacological, and lifestyle modification therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 and above
* Systolic BP ranging from 130-139mmHg and/or diastolic BP ranging from 80-89mmHg

Exclusion Criteria:

* Unable, unwilling, or incompetent to provide informed consent
* Physically unable to come to the study visits, or to sit comfortably in a chair for up to two hours at a time
* Weight is over the chair limit (285 pounds)
* Known atherosclerotic cardiovascular disease
* Cardiovascular risk score of ≥ 10% (per http://tools.acc.org/ASCVD-Risk-Estimator-Plus/#!/calculate/estimate/)
* Prior diagnosis of stage 2 hypertension
* Ongoing need for treatment of hypertension with medications
* Known seizure disorder
* Known or anticipated pregnancy
* Severe hearing impairment (because the subject will be using headphones during the interventions)
* Ongoing need for treatment with opiate, benzodiazepine, or anti-psychotic medications, anti-depressant medications such as SSRI, SNRI, or tricyclic, and sleep medications such as zolpidem or eszopiclone
* Anticipated and ongoing use of recreational drugs, alcohol, or energy drinks
* Ongoing need for treatment with thyroid medications
* Are enrolled in another research study that includes an active intervention
* Have previously received brainwave optimization (BWO), used a B2 or B2v2 wearable device, or previously participated in a HIRREM research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Tegeler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Department of Neurology, Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIRREM | Continued Current Care
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIRREM | Continued Current Care | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.00 (1.41) | 68.33 (15.50) | 54.60 (21.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Blood Pressure, as Measured by an Automated Oscillometric Blood Pressure Device.
Description: BP will be obtained in the left arm, with the participant sitting comfortably, and the left arm resting on a desk/table. Three samples will be obtained and the last two averaged to get the value that will be used as the reading. Primary outcome will be at V3 (4-6 weeks post final session).
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
mmHg
  ∆_V1_V3 Systolic | -3.00 (8.49) | -6.67 (22.55)
  ∆_V1_V3 Diastolic | -6.00 (4.24) | -7.67 (13.80)

2. Secondary Outcome: Change in Heart Rate Variability (SDNN)
Description: Heart rate variability is measured in the time domain as standard deviation of beat-to-beat interval
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
ms | 17.55 (16.48) | 9.47 (3.83)

3. Secondary Outcome: Change in Baroreflex Sensitivity
Description: Blood pressure and heart rate are acquired from 10 minute recordings of noninvasive finger arterial pressure measurements and ECG with participants lying quietly, supine. Systolic BP and beat to beat, RR intervals files generated via the data acquisition system at 1000 Hz, are analyzed using Nevrokard BRS software. Analysis is conducted on the first complete 5-minute epoch. Power spectral densities of systolic blood pressure (SBP) and R-R interval (RRI) oscillations are computed by 512 points Fast Fourier Transform (FFT) and integrated over specified frequency ranges (HF: 0.15-0.4 Hz). The square-root of the ratio of RRI's and SBP powers is computed to calculate HF alpha indices, which reflect BRS. The software scans the RRI and SBP records, identifies sequences, and calculates linear correlation between RRI and SBP for each sequence. A measure of sequence BRS is then calculated as Sequence ALL.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
ms/mmHg | 0.35 (12.66) | -4.97 (28.14)

4. Secondary Outcome: Change in Insomnia Severity Index (ISI)
Description: The severity of insomnia symptoms is measured using the ISI with each data collection visit. The ISI is a 7 question measure, with responses from 0-4 for each question, yielding scores ranging from 0-28. Higher scores indicate the strength of the insomnia severity.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
score on a scale | -3.00 (2.83) | -2.67 (5.13)

5. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI is a 19 item inventory that assesses sleep quality over a 1-month time interval. Items are weighted on a 0-3 interval scale. A global PSQI score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
score on a scale | 0 (1.41) | -1.33 (1.53)

6. Secondary Outcome: Change in Epworth Sleepiness Score (ESS)
Description: The ESS measures a person's general level of daytime sleepiness, or their average sleep propensity in daily life. The simple questionnaire is based on retrospective reports of the likelihood of dozing off or falling asleep in a variety of different situations. Rated on a 4-point scale (0-3), it evaluates their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. Lower scores denote a lower level of daytime sleepiness.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
score on a scale | 1.50 (2.12) | -0.67 (2.08)

7. Secondary Outcome: Change in Center for Epidemiologic Studies Depression Scale (CES-D)
Description: The CES-D is a 20-item survey assessing affective depressive symptomatology to screen for risk of depression. Scores range from 0-60, with a score of 16 commonly used as a clinically relevant cut-off. Higher scores indicate the presence of more symptomatology.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
score on a scale | 7.00 (1.41) | 1.33 (5.13)

8. Secondary Outcome: Change in Generalized Anxiety Disorder-7 (GAD-7)
Description: The GAD-7 is a seven item screening tool for anxiety that is widely used in primary care. Scores range from 0-21. A lower score denotes a lower level of anxiety.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
score on a scale | 4.50 (3.54) | 1.00 (1.00)

9. Secondary Outcome: Change in PTSD Checklist for Civilians (PCL-C)
Description: The PCL-C measures the American Psychiatric Association's Diagnostic and statistical manual of mental disorders (DSM-IV) Criteria B, C, & D of PTSD symptoms based on traumatic life experience related to civilians. Seventeen items are rated on a Likert scale with a composite score range of 17 to 85. A score of 44 or higher correlates with probability of civilian-related PTSD.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
score on a scale | 6.00 (9.90) | -4.00 (5.20)

10. Secondary Outcome: Change in Perceived Stress Scale (PSS)
Description: The PSS is a ten-item psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Scores range from 0-40. A lower score denotes a lower level of perceived stress.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
score on a scale | 5.50 (4.95) | -3.33 (1.15)

11. Secondary Outcome: Change in International Physical Activity Questionnaire (IPAQ-SF)
Description: This is a four item questionnaire asking about physical activity in the last 7 days. Scores are calculated and categorized as low, moderate, or high. A higher score denotes more physical activity. For results, categories could not be presented so they were coded as: 1=low, 2=moderate, and 3=high.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
score on a scale | 0.00 (2.83) | 0.00 (0.00)

12. Secondary Outcome: Change in HIRREM Physical Activity Satisfaction Questions
Description: This is a four item questionnaire asking about the participants level of satisfaction with their physical activity. Responses range from 0-6 for each question, yielding scores ranging from 0-24. Higher scores denote a higher level of satisfaction.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
score on a scale | 3.50 (2.12) | 2.00 (3.46)

13. Secondary Outcome: Change in Quality of Life Scale (QOLS)
Description: The QOLS ) is a 16-item scale that was modified from a 15-item scale used in chronic disease patients. Topics include different components of daily life such as relationships, community engagement, personal fulfillment, and recreation. Each item is scaled from 1 to 7 and a sum score is calculated to represent higher levels of satisfaction in life (range is 16-112).
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
score on a scale | -4.00 (5.66) | 4.33 (7.23)

14. Secondary Outcome: Change in Drop Stick Reaction Time
Description: Reaction testing will be evaluated by a drop-stick, clinical reaction time apparatus. The apparatus is placed between the thumb and index finger of the subject and released at a random time during a countdown. The subject catches the apparatus and the distance fallen (cm) is converted to reaction. Following two practice trials, participants perform eight trials, and a mean distance value is calculated. This is repeated with a second set of 8 trials later during the enrollment visit, and the mean distance value from the second trial will be used as the baseline value. Use of the average distance from the second set of trials will be used as the baseline value so as to avoid the impact of learning effect for this test. Only one set of trials will be used for comparison at follow up data collections. A lower average indicates a faster reaction time.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
cm | -0.06 (0.27) | -0.96 (3.01)

15. Secondary Outcome: Change in Grip Strength
Description: Grip strength will be evaluated using a hydraulic hand dynamometer (Baseline Hydraulic Hand Dynamometer). Participants will squeeze the dynamometer three times in each hand. The scores from each hand will be averaged separately. A higher score indicates stronger grip strength.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
lbs
  ∆_V1_V3 Right Hand | 16.17 (18.15) | 0.00 (6.01)
  ∆_V1_V3 Left Hand | -2.33 (3.77) | 2.44 (5.54)

16. Other Pre Specified Outcome: Change in Alcohol Intake Screening (Audit-C)
Description: The AUDIT-C is a short, 3-item alcohol screening for hazardous drinkers or active alcohol use disorders. This measure consists of 3 questions to assess an individual's alcohol use. Each question has five possible answers ranging from of 0-4 with a total scoring scale of 0-12. A total score of three or more in women and a score of four or more in men is suggestive of hazardous drinking or active alcohol use disorders.
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM | Continued Current Care
Number analyzed (Participants) | 2 | 3
score on a scale | -1.50 (0.71) | 0.00 (0.00)

ADVERSE EVENTS:
Time Frame: Baseline to V3 (4-6 weeks following completion of the intervention for HCC, 8-10 weeks after V1 for CCC).
Arm/Group | HIRREM | Continued Current Care
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

LIMITATIONS AND CAVEATS:
We found that the blood pressure requirements and medication exclusions we originally set in place were very hard to meet and therefore, excluded many subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT03479697/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT03479697/ICF_001.pdf